CLINICAL TRIAL: NCT01813994
Title: Role of Statin on the Gastric Inflammation in Patients at High Risk of Gastric Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4-2012-0889
Record Dates: First submitted 2013-03-07; First posted 2013-03-19 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2018-12

CONDITIONS: Early Gastric Cancer or Gastric Adenoma
Keywords: Statin; Gastric inflammation; Gastric cancer
MeSH Terms: conditions — Stomach Neoplasms; Gastritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Placebo Comparator): Without simvastatin
  Interventions: Drug: Arm2: Placebo
- Statin group (Experimental): With simvastatin
  Interventions: Drug: Arm1: Statin

INTERVENTIONS:
Drug: Arm1: Statin — Study1 (only H. pylori infected patients) Arm1: All patients undergo H. pylori eradication therapy after 2 weeks from the endoscopic submucosal dissection. In this arm2, all patients take statins for 6 months. Then, follow-up endoscopy for gastric biopsy and CLO test will be performed after 6.5 months from the endoscopic submucosal dissection.
  Study2 (only H. pylori non-infected patients) Arm1: In this arm2, all patients start taking statins after 2 weeks from the endoscopic submucosal dissection. Follow-up endoscopy for gastric biopsy will be performed after 6.5 months from the endoscopic submucosal dissection.
  Arms: Statin group
Drug: Arm2: Placebo — Study1 (only H. pylori infected patients) Arm2: All patients undergo H. pylori eradication therapy after 2 weeks from the endoscopic submucosal dissection. In this arm2, all patients take placebos for 6 months. Then, follow-up endoscopy for gastric biopsy and CLO test will be performed after 6.5 months from the endoscopic submucosal dissection.
  Study2 (only H. pylori non-infected patients) Arm2: In this arm2, all patients start taking placebos after 2 weeks from the endoscopic submucosal dissection. Follow-up endoscopy for gastric biopsy will be performed after 6.5 months from the endoscopic submucosal dissection.
  Other Names: C10AA-Hmg coa reductase inhibitors
  Arms: Control group

SUMMARY:
Statins are commonly used as cholesterol-lowering medications and have shown effectiveness in the primary and secondary prevention of heart attack and stroke. In addition, several recent studies of human cancer cell lines and animal tumor models indicate that statins may have chemopreventive properties through the arresting of cell-cycle progression. The chemopreventive effect of statins was demonstrated in some kind of human tumors including colorectal cancer. In addition, recent one large epidemiologic study showed that statins decreased risk of gastric cancer. On the other hands, it has been well known that Helicobacter pylori infection induces gastric atrophy and intestinal metaplasia, which are premalignant lesions of gastric cancer. Progression of these premalignant lesions could be limited by H. pylori eradication. In addition, a recent double blind randomization study revealed that simvastatin as adjuvant to standard therapy improves significantly the H. pylori eradication rate. Therefore, investigators conjecture that statins may have an adjuvant role for inhibition of gastric carcinogenesis. investigators aim to evaluate the role of statins in gastric carcinogenesis by observing the changes of gastric inflammation under statins.

ELIGIBILITY:
Inclusion Criteria:

1. Age, between 20 and 70
2. Early gastric cancer or adenoma which is achieved curative resection by endoscopic submucosal dissection
3. ECOG performance status 0 or 1

Exclusion Criteria:

1. Previous subtotal gastrectomy or gastrostomy
2. Repeated endoscopic submucosal dissection
3. Two or more synchronous lesions
4. Presence of gastric or duodenal ulcer except artificial ulcer due to endoscopic submucosal dissection
5. History of drugs which are able to induce gastric ulcer including aspirin, NSAIDs, and steroid (30 days or more, within 1 year at the time of screening
6. Indication of statins, including dyslipidemia, myocardial infarction, and heart failure.
7. Develop of complications caused by endoscopic submucosal dissection, including bleeding, perforation, and pneumonia
8. LDL < 70 mg/dL
9. Allergy to statins
10. Pregnancy or breast milk feeding
11. Active infection
12. Significant cardiopulmonary disease
13. Active hepatitis or severe hepatic dysfunction
14. Severe renal dysfunction
15. Severe bone marrow dysfunction

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2014-11; Primary Completion 2018-06-19 (Actual); Study Completion 2018-06-19 (Actual)

PRIMARY OUTCOMES:
Proportion of the patients with high-risk (III/IV) OLGA stages | 6 months from the start of taking the statins
  patients with high-risk OLGA stages will be assessed by histologic examinations

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea